CLINICAL TRIAL: NCT05509530
Title: Efficacy and Safety Study of Anti-BCMA/GPRC5D CAR-T Cells in Subjects With Relapsed and Refractory Multiple Myeloma
Brief Title: Safety and Efficacy of Anti-BCMA/GPRC5D CAR-T Cell Therapy in Treating Relapsed and Refractory Multiple Myeloma(rr/MM)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Kai Lin Xu，MD, Principal Investigator, Xuzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XYFY2022-KL118-01
Record Dates: First submitted 2022-08-02; First posted 2022-08-22 (Actual); Last update posted 2022-08-22 (Actual); Status verified 2022-08

CONDITIONS: Multiple Myeloma
Keywords: Multiple Myeloma; BCMA; GPRC5D
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti BCMA/GPRC5D CAR-T (Experimental): Enrolled patients will receive prespecified dose of autologous anti BCMA/GPRC5D CAR-T cells.
  Interventions: Other: anti-BCMA/GPRC5D CAR-T CELL

INTERVENTIONS:
Other: anti-BCMA/GPRC5D CAR-T CELL — anti-BCMA/GPRC5D autologous CAR T cells will be infused at a dose ranging from 1 - 2 x 10^6/kg CAR+ T cells after receiving lymphodepleting chemotherapy

SUMMARY:
This is an open label, single-arm, Phase 2 study to evaluate the efficacy and safety of Anti-BCMA/GPRC5D CAR-T in subjects with relapsed and refractory multiple myeloma. A leukapheresis procedure will be performed to manufacture Anti-BCMA/GPRC5D chimeric antigen receptor (CAR) modified T cells. Prior to Anti-BCMA/GPRC5D infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide.

DETAILED DESCRIPTION:
This open label, single-arm, Phase 2 study aims to evaluate the efficacy and safety of Anti-BCMA/GPRC5D CAR-T in subjects with relapsed and refractory multiple myeloma. A leukapheresis procedure will be performed to manufacture Anti-BCMA/GPRC5D chimeric antigen receptor (CAR) modified T cells. Prior to Anti-BCMA/GPRC5D infusion subjects will receive lymphodepleting therapy with fludarabine and cyclophosphamide. After infusion, the investigators will observe the characteristics of dose limited toxicity (DLT), and determine the maximum tolerable agent MTD and rp2d were confirmed. To provide basis for the dosage and treatment plan of cell products in follow-up clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Age and gender: 18 years old <= age <= 70 years old, gender unlimited, signing informed consent voluntarily;
2. According to the classification definition of IMWG standard, the diagnosis of plasmacytoma is multiple myeloma, plasmacytic leukemia, poems syndrome, monoclonal IMMUNOGLOBULINEMIA, primary macroglobulinemia or primary amyloidosis which are invalid or relapsed after at least three-line treatment (including chemotherapy based on bortezomib and / or lenalidomide);
3. BCMA and GPRC5D were positive on the surface of plasma membrane;
4. The patients could not receive the treatment of HSCT, or the relapse after HSCT was judged to need treatment by researchers;
5. ECOG score is 0 or 1;
6. Expected survival time >= 12 weeks;
7. The subjects must have proper organ function and meet all the following laboratory test results before entering the group

   1. Blood routine test: neutrophil >= 1.0 x 10^9 / L; hemoglobin >= 70 g / L; platelet >= 50 x 10^9 / L;
   2. Liver function: ALT and AST <= 2.5 x ULN; total bilirubin <= 1.5 x ULN;
   3. Renal function: serum creatinine <= 2.5 x ULN; or creatinine clearance calculated according to Cockcroft Gault formula Rate CrCl >= 60 ml / min.
   4. Electrolyte: blood potassium >= 3.0 mmol / L; blood calcium >= 2.0 mmol / L; blood magnesium >= 0.5 mmol / L;
   5. Coagulation function: fibrinogen >= 1.0g/l; activated partial thromboplastin time (APTT) <= Keywords ULN + 10s; prothrombin time (PT) < ULN + 3S;
8. The subjects should be willing to provide effective diagnosis evidence or bone marrow examination before treatment, and bone marrow or effective examination after treatment;
9. Women of childbearing age and fertile male subjects must take one of the following effective contraceptive measures from signing informed consent until one year after anti-BCMA/GPRC5D CAR-T cell transfusion: abstinence, double barrier contraceptive method, IUD, hormone contraceptive;
10. Male subjects were forbidden to donate sperm from signing the informed consent until one year after anti-BCMA/GPRC5D CAR-T cell transfusion;
11. Sign informed consent

    1. The subject must have informed consent to the test before the test, and be voluntary by himself (or his legal representative) signed the written informed consent;
    2. The subjects or their legal representatives can communicate well with the researchers and follow the protocol to complete the test.

Exclusion Criteria:

1. Previous treatment history

   1. Received hematopoietic stem cell transplantation within 2 months before the start of administration, or within the screening period after transplantation, immunosuppressive therapy was used because of graft-versus-host disease;
   2. Patients who had received chemotherapy, immunotherapy, radiotherapy and major surgery within 4 weeks before the start of administration;
   3. Those who received the live vaccine within 4 weeks before the start of administration and / or planned to receive the live vaccine after the trial;
   4. Those who have received clinical trial drug treatment or are participating in other clinical trials within 4 weeks before drug administration;
2. History of disease and operation

   1. Patients with central nervous system invasion by plasmacytoma;
   2. Hypertension and drug treatment can not get good control (blood pressure > 140 / 90 mmHg);
   3. Doppler ultrasound evaluation: left ventricular ejection fraction (LVEF) < 50%;
   4. Arrhythmia with NCI CTCAE 5.0 grade >= 2, or male QTc > 450 ms, female QTc > 470 MS (QTc was calculated by the friderica correction formula QTc = QT / rr0.33); patients with a history of tip torsion or congenital QT prolongation syndrome;
   5. Patients with any of the following diseases within 12 months before administration: myocardial infarction, severe or unstable heart, patients with colic, coronary artery bypass or peripheral artery bypass grafting, congestive heart failure, cerebrovascular events (including transient ischemic attack), etc;
   6. During the screening period, the researchers judged that there were uncontrollable and active infectious diseases;
   7. People infected with human immunodeficiency virus (HIV);
   8. HBsAg was positive and in the active phase of hepatitis B (HBV DNA quantity >= 1.00 x 10^2 copies / ml);
   9. Hepatitis C antibody (anti HCV) was positive and was in the active phase of hepatitis C (hepatitis C RNA was not in the normal mode)Perimetric value);
   10. The researchers judged patients with severe electrolyte disorder;
   11. Patients with a clear tendency of gastrointestinal bleeding, including the following: local active ulcer focus, and stool occult blood (>= + +); patients with a history of black stool and hematemesis within 2 months; researchers believe that digestion may occur Patients with massive bleeding of the Tao;
   12. Patients with a history of solid organ transplantation;
   13. The investigator or sponsor thinks that he / she has other acute, serious or chronic medical or psychological diseases and is not suitable for participation Add clinical trial;
   14. Pregnant and nursing women
3. Prohibited treatment and / or medication

   1. At the same time, other anti-tumor drugs, including traditional Chinese medicine, were used;
   2. At the same time, take drugs that can prolong QT interval (including class IA and III antiarrhythmic drugs);
   3. Those who need to receive oxygen every day;
   4. Long term use of corticosteroids (except for local inhalation);
4. others

   1. Those who have a history of psychoactive drug abuse and are unable to give up or have mental disorders;
   2. Habitually drink grapefruit juice or excessive tea, coffee and / or caffeinated beverages during the trial Unable to give up;
   3. According to the judgment of the researchers, there are serious concomitant diseases endangering the safety of patients or affecting the completion of the trialillnes.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Adverse Events, with abnormal vital signs, abnormal physical examination findings, abnormal laboratory test results, abnormal ECGs and abnormal echocardiograms. | 12 months

SECONDARY OUTCOMES:
overall response rate (ORR) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for MM | 24 months
  Percentage of subjects who achieved a CR, VGR, PR according to IMWG Uniform Response Criteria for Multiple Myeloma (MM)
complete response (CR) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for MM | 24 months
  Percentage of subjects who achieved a CR according to IMWG Uniform Response Criteria for Multiple Myeloma (MM)
very good partial response (VGPR) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for MM | 24 months
  Percentage of subjects who achieved a VGPR according to IMWG Uniform Response Criteria for Multiple Myeloma (MM)
partial response (PR) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for MM | 24 months
  Percentage of subjects who achieved a PR according to IMWG Uniform Response Criteria for Multiple Myeloma (MM)

CONTACTS AND LOCATIONS:
Overall Officials: Kailin Xu, M.D., Ph.D., Principal Investigator — Xuzhou Medical University
Locations (1):
- Kailin Xu, Xuzhou, Jiangsu, China

REFERENCES:
- [Derived] Zhou D, Sun Q, Xia J, Gu W, Qian J, Zhuang W, Yan Z, Cheng H, Chen W, Zhu F, Qi K, Li D, Sang W, Zhu L, Ma S, Li H, Zhang H, Qiu T, Yan D, Zhang Y, Peng S, Chang AH, Xu K, Li Z. Anti-BCMA/GPRC5D bispecific CAR T cells in patients with relapsed or refractory multiple myeloma: a single-arm, single-centre, phase 1 trial. Lancet Haematol. 2024 Oct;11(10):e751-e760. doi: 10.1016/S2352-3026(24)00176-5. Epub 2024 Jul 23. PMID 39059405